CLINICAL TRIAL: NCT03248544
Title: Effect of Single High Dose Vitamin D3 on Peri-operative and Post-operative Complications and Clinical Outcomes in Patients Under Craniotomy for Brain Tumor Resection
Brief Title: Therapeutic Benefit of Preoperative Supplemental Vitamin D in Patients Undergoing Brain Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1396-607
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Brain Neoplasms
Keywords: vitamin D; Brain Neoplasms; perioperative complications; clinical outcomes; craniotomy; Immune System
MeSH Terms: conditions — Brain Neoplasms | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D (Experimental): Intervention patients will be received a single dose of 300000 IU vitamin D via intramuscular injection
  Interventions: Drug: vitamin D
- control (Other): Control patients will not be received any intervention
  Interventions: Other: control

INTERVENTIONS:
Drug: vitamin D — Fat-soluble vitamin D injection contain of 300,000 IU vitamin D that given via intramuscular injection
  Other Names: Cholecalciferol
  Arms: vitamin D
Other: control — No intervention
  Arms: control

SUMMARY:
Vitamin D supplementation not only has beneficial effects on morbidity and mortality in critically ill patients but it may also lead to alleviate of seizure, brain edema, infection, pain and some other perioperative complications, possibly in part through an attenuation of the immune response.In this trial patients with brain tumor under craniotomy will receive a single high dose vitamin D compared to control group.

DETAILED DESCRIPTION:
A randomized, double blind, controlled trial will be conducted in neurosurgery ward, operating room (OR) and intensive care unit (ICU) in Tehran, Iran. After a full review of the inclusion and exclusion criteria and explanation of the risks and benefits of the study, written consent form will be completed. The participants are 60 eligible hospitalized patients that diagnosed with brain tumor and need to craniotomy, aged ≥ 18 years. Intervention patients will be received an intramuscular (IM) single dose of vitamin D (300000 IU). Patients will be evaluated for occurrence of perioperative complications and clinical outcomes immediately after surgery until 1 month later and 1 and 6 months mortality.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of patient or legal representative
* 25(OH)D level below 20ng/dL

Exclusion Criteria:

* Other trial participation, including previous participation in the pilot trial
* Pregnant or lactating women
* Hypercalcemia
* Hyperphosphatemia
* Tuberculosis
* Sarcoidosis
* History of nephrolithiasis
* History of hyperparathyroidis
* Medications that interfere with vitamin D metabolism
* Renal Insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D level | Postoperative day 5
  25(OH) will be measured after surgery

SECONDARY OUTCOMES:
Peri-operative Complications | During surgery, recovery and hospitalization (5 days post op)
  Complications in operating room, recovery room, ICU and neurosurgery ward
Post-operative Complications | 30 days after surgery
  Complications after hospital discharge
Duration of stay in ICU | 30 days
  Length of stay in ICU is measured
Duration of stay in hospital | 30 days
  Length of stay in hospital is measured
1-month mortality | 30 days
  Mortality during hospitalization or 1 month after surgery
6-month mortality | 6 months
  Mortality during 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, PhD, Study Chair — Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (2):
- Iran (2):
  - Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran
  - Shohada Tajrish Hospital, Tehran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hajimohammadebrahim-Ketabforoush M, Shahmohammadi M, Keikhaee M, Eslamian G, Vahdat Shariatpanahi Z. Single high-dose vitamin D3 injection and clinical outcomes in brain tumor resection: A randomized, controlled clinical trial. Clin Nutr ESPEN. 2021 Feb;41:153-159. doi: 10.1016/j.clnesp.2020.11.027. Epub 2021 Jan 2. PMID 33487259